CLINICAL TRIAL: NCT06393426
Title: The Constitution and Efficacy of Chinese Medicine of Infertility Male and Female, and Pregnant Female: a Retrospective Study
Brief Title: The Constitution and Efficacy of Chinese Medicine of Infertility Male, Female, and Pregnant Female
Status: Completed | Type: Observational
Sponsor: China Medical University Hospital (Other)
Responsible Party: Principal Investigator, Shan-Yu Su, Attending Physician, Traditional Chinese Medicine Obstetrics and Gynecology, China Medical University Hospital
Other Study IDs: CMUH111-REC2-085
Record Dates: First submitted 2024-04-06; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Infertility; Miscarriage Threatening
Keywords: infertility; Chinese Medicine; miscarriage prevention; retrospective study
MeSH Terms: conditions — Infertility; Abortion, Threatened | interventions — Ephedrae herba

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Chinese Herb — Chinese herbal medicine

SUMMARY:
The project aims to conduct a retrospective study to assess the impact of Traditional Chinese Medicine (TCM) on improving pregnancy rates and preventing miscarriages. It will include patients with infertility issues or a history of miscarriage. The study will analyze demographic and physiological data, TCM constitution, basal body temperature, reproductive history for females, and semen analysis for males, to determine the effectiveness of TCM care in enhancing fertility outcomes.

DETAILED DESCRIPTION:
The present project plans to conduct a retrospective study based on the data of the National Health Insurance Traditional Chinese Medicine Enhancement Quality of Maternity Care Plan.

Analysis Methods: The collected data was archived using SPSS software, and the following testing methods were employed for statistical analysis among different datasets:

1. Paired-t Test: Examining differences in temperature and duration between follicular and luteal phases in females before and after treatment.
2. Chi-Square Test: Assessing the relationship between traditional Chinese medicine constitution and pregnancy outcomes.
3. McNemar Test: Testing the significance of changes in traditional Chinese medicine constitution before and after treatment.
4. Logistic Regression: Conducting multivariate analysis to explore factors associated with pregnancy status.

The purpose of this project is to figure out after conducting proper Chinese medical care, whether it will improve the target patients' pregnancy rate and miscarriage prevention rate. Those data will conduct a biological analysis to compare the difference between pregnancy and miscarriage prevention rates between different patients.

ELIGIBILITY:
Inclusion Criteria:

* Fertility Assistance: For male and female patients who have been married for over a year with regular sexual activity but are unable to conceive.
* Miscarriage Prevention: For females who have had miscarriages, non-natural conception, conception through fertility assistance, and are prone to miscarriage.

Exclusion Criteria:

* Fertility Assistance:

  1. Incomplete demographic data for males/females
  2. Incomplete Traditional Chinese Medicine constitution determination data for males/females
  3. Incomplete information on the follicular/luteal phase for females
  4. Incomplete semen analysis data for males
* Miscarriage Prevention:

  1. Incomplete demographic data
  2. Incomplete physiological examination data
  3. Incomplete data on related disease records

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients who met the following criteria, from 2015 to 2020, were reported by various medical institutions across Taiwan into the National Health Insurance database for the Traditional Chinese Medicine Enhancement of Maternity Care Quality Project.
Sampling Method: Non-Probability Sample
Enrollment: 37611 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-05-31 (Actual)

PRIMARY OUTCOMES:
Temperature of follicular phase | through study completion, an average of 254 days
  To determine whether there is a difference in the temperature of the follicular phase
Days of follicular phase | through study completion, an average of 254 days
  To determine whether there is a difference in the days of the follicular phase
Temperature of luteal phase | through study completion, an average of 254 days
  To determine whether there is a difference in the temperature of the luteal phase
Days of luteal phase | through study completion, an average of 254 days
  To determine whether there is a difference in the days of the luteal phase

SECONDARY OUTCOMES:
TCM constitution and pregnancy | through study completion, an average of 254 days
  To detect the correlation between TCM constitution and pregnancy

CONTACTS AND LOCATIONS:
Locations (1):
- CMUH, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No